CLINICAL TRIAL: NCT00554827
Title: A Phase 1, Open-label Study of Pralatrexate With Vitamin B12 and Folic Acid Supplementation in Patients With Relapsed or Refractory Cutaneous T-cell Lymphoma
Brief Title: Study of Pralatrexate in Patients With Relapsed or Refractory Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-010
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: Relapsed or Refractory Cutaneous T-cell Lymphoma; Lymphoma; Cutaneous T-cell Lymphoma; T-cell Lymphoma; Mycosis fungoides; Sézary syndrome; Primary cutaneous anaplastic large cell
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Recurrence; Lymphoma; Lymphoma, T-Cell; Mycosis Fungoides; Sezary Syndrome | interventions — Vitamin B 12; Folic Acid; 10-propargyl-10-deazaaminopterin

ARMS (1):
- Pralatrexate Injection (FOLOTYN,PDX,Pralatrexate(R (Experimental): Intravenous (IV) push over 3-5 minutes into a patent IV line containing normal saline (0.9% sodium chloride).
  Pralatrexate will be administered via intravenous (IV) push over 3-5 minutes. The frequency of pralatrexate will be administered weekly for 3 or 4 weeks (depending on cohort), with 1 week of rest.
  Interventions: Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid; Drug: Pralatrexate

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — 1 mg intramuscular injection
  Administered at least 10 days prior to start of pralatrexate if patient has elevated methylmalonic acid (MMA) and/or homocysteine(Hcy) levels.
  Administered every 8-10 weeks throughout the study and for at least 30 days after last dose of pralatrexate.
  Other Names: Cyanocobalamin
Dietary Supplement: Folic Acid — 1 mg orally
  Administered at least 10 days prior to start of pralatrexate if patient has elevated methylmalonic acid (MMA) and/or homocysteine(Hcy) levels.
  Administered daily throughout the study and for at least 30 days after last dose of pralatrexate.
  Other Names: Vitamin B9; Folate; Folacin
Drug: Pralatrexate — Intravenous (IV) push over 3-5 minutes into a patent IV line containing normal saline (0.9% sodium chloride). Pralatrexate will be administered via intravenous (IV) push over 3-5 minutes. The frequency of pralatrexate will be administered weekly for 3 or
  Other Names: FOLOTYN,PDX,Pralatrexate,(RS)-10-propargyl-10-deazaaminopterin

SUMMARY:
This study is being conducted to identify how much and how often pralatrexate, given with vitamin B12 and folic acid, can be given safely to patients with cutaneous T-cell lymphoma (CTCL) that has relapsed (returned after responding to previous treatment) or is refractory (has not responded to previous treatment). It is also being conducted to get information on whether or not pralatrexate is effective in treating relapsed or refractory CTCL.

DETAILED DESCRIPTION:
This is a Phase 1, single-arm, open-label, multi-center study designed to determine an effective and well-tolerated dose and schedule of pralatrexate when administered concurrently with vitamin B12 and folic acid supplementation to patients with relapsed or refractory CTCL. The start of study treatment is defined as the initiation of pralatrexate. A patient may begin pralatrexate, provided he/she has methylmalonic acid (MMA) serum concentrations < 200 nmol/L and homocysteine (Hcy) concentrations < 10 μmol/L at screening. If a patient has elevated MMA and/or Hcy concentrations, vitamin supplementation will be initiated at least 10 days prior to pralatrexate initiation. Once the patient is on study, the dosing of vitamin supplementation must adhere to the schedule defined by the protocol. Vitamin supplementation will consist of vitamin BB12

1 mg intramuscular (IM) every (q) 8-10 weeks, and folic acid 1 mg by mouth (PO) once a day (QD).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed relapsed or refractory cutaneous T-cell lymphoma (CTCL):

  1. Mycosis fungoides Stage IB or higher
  2. Sézary syndrome
  3. Primary cutaneous anaplastic large cell
* No curative treatment options.
* Progression of disease (PD) or relapse of disease after at least 1 previous systemic therapy, PD after last prior treatment regimen, and recovered from the toxic effects of prior therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Life expectancy ≥ 3 months.
* Adequate blood, liver, and kidney function as determined by laboratory tests.
* Methylmalonic acide (MMA) serum concentration < 200 nmol/L and homocysteine (Hcy) concentration < 10 μmol/L at screening, or receipt of 1 mg daily oral folic acid for at least 10 days prior to the planned start of pralatrexate and 1 mg intramuscular vitamin B12 within 10 weeks of the planned start of pralatrexate.
* Women of childbearing potential must use a medically acceptable contraceptive regimen from study treatment initiation until at least 30 days after the last dose of pralatrexate and must have a negative serum pregnancy test within 14 days prior to the first day of study treatment. Serum pregnancy test not required for patients who are postmenopausal (greater than 12 months since last menses) or are surgically sterilized.
* Women who are breastfeeding.
* Men who are not surgically sterile must use a medically acceptable contraceptive regimen from start of pralatrexate until at least 90 days after the last administration of pralatrexate.
* Written informed consent and privacy authorization.

Exclusion Criteria:

* Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy, the patient must be disease-free for ≥ 5 years. Patients with other prior malignancies < 5 years before study entry may be enrolled if treatment resulted in complete resolution of the cancer and currently have no clinical, radiologic, or laboratory evidence of active or recurrent disease.
* Congestive heart failure Class III/IV per the New York Heart Association Heart Failure Guidelines.
* Uncontrolled hypertension.
* Human immunodeficiency virus (HIV)-positive diagnosis with a CD4 count of <100 mm3 or detectable viral load within the past 3 months, and is receiving combination anti-retroviral therapy.
* Symptomatic central nervous system metastases or lesions for which treatment is required.
* Active uncontrolled infection, underlying medical condition that would impair ability to receive protocol treatment.
* Major surgery within 2 weeks of planned start of treatment.
* Receipt of any conventional chemotherapy or radiation therapy (RT) encompassing >10% of bone marrow within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study treatment or planned use during the study.
* Receipt of systemic corticosteroids within 3 weeks of study treatment, unless on a continuous dose of ≤10 mg/day of prednisone for at least 1 month.
* Initiation of or change in dosage of topical corticosteroids within 3 weeks of study treatment (topical steroid use within 3 weeks is allowed if strength/use has been stable for at least 1 month; topical corticosteroids cannot be started during the study).
* Use of investigational drugs, biologics, or devices within 4 weeks prior to study treatment or planned use during the study.
* Receipt of a monoclonal antibody within 3 months without evidence of progression.
* Use of oral retinoids within 4 weeks of study treatment or high-dose vitamin A.
* Previous exposure to pralatrexate, unless the patient was on this study, achieved a complete or partial response, and was taken off study treatment because of investigator decision, and subsequently experienced disease recurrence or progressive disease.
* Re-entering patients: must not have received subsequent therapy for CTCL during the time off initial study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-08; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Determine an Effective and Well-tolerated Dose and Schedule of Pralatrexate with Vitamin B12 and Folic Acid Supplementation for Patients with Relapsed or Refractory Cutaneous T-cell Lymphoma (CTCL) | Assessed at the end of every even-numbered cycle (every 8 weeks) for the first 6 months, then every 4 cycles (16 weeks)
  Response rate was used as the primary measure of efficacy during the process of identifying a well-tolerated and effective dosing regimen of pralatrexate in patients with relapsed/refractory CTCL. Duration of response was defined as the number of days between the date of first tumor response assessment of objective response (CR, CRu, or PR, whichever was recorded first) and the first date that recurrent disease or PD was objectively documented or death.

SECONDARY OUTCOMES:
Characterize the Safety Profile of Pralatrexate in Patients with Relapsed or Refractory CTCL. | Assessed at all study visits: weekly while on treatment and at safety follow-up (35 +/- 5 days post-last dose) or early termination visit (at time of withdrawal)
  The safety analysis set included all patients who received at least 1 dose of pralatrexate. In order to be considered evaluable in the dose-finding phase of the study, patients must have
  (a) either experienced a DLT or (b) received all planned doses within the first cycle. Patients who terminated from the study prior to completion of cycle 1 for reasons other than DLTs were replaced.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saunders, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (10):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - Stanford University School of Medicine, Redwood City, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington